CLINICAL TRIAL: NCT00157638
Title: Optimizing Drug Therapy in Primary Care: Integrating Pharmacists With Ontario Family Physician Group Practices.
Brief Title: Integrating Family Medicine and Pharmacy to Advance Primary Care Therapeutics
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Organization: McMaster University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: G03-02671
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2006-09-11 (Estimated); Status verified 2006-09

CONDITIONS: Diabetes; Hypertension; Hyperlipidemia; Constipation; Pain
Keywords: pharmacist; physician; primary care; collaboration; therapeutics
MeSH Terms: conditions — Diabetes Mellitus; Hypertension; Hyperlipidemias; Constipation; Pain

INTERVENTIONS:
Behavioral: integration of pharmacist into primary care
Drug: optimizing therapeutic treatments
Behavioral: optimizing processes of care

SUMMARY:
Recent health policy documents have endorsed an integrated model of collaboration between pharmacists and physicians in primary care. The integration of pharmacists into primary care has been identified as a priority for primary health care reform in Canada. However, the best way to do this has not been demonstrated or evaluated. This demonstration project shows the various ways in which pharmacists can be trained and integrated into different family practice settings, the processes and costs associated with doing this, and the outcomes observed. The main hypothesis is that pharmacist integration into family practice will optimize medication use, clinical care and clinical outcomes. This information provides policy makers with necessary information about collaboration between pharmacists and family physicians for their overall goal of reforming the delivery of primary health care to the population.

DETAILED DESCRIPTION:
The overall goal of IMPACT was to improve patient outcomes by optimizing drug therapy through a community practice model that integrates pharmacists into family practices.

This multi-site demonstration project involved 7 pharmacists, approximately 70 physicians and approximately 150,000 patients. Within each practice site, a pharmacist with special clinical training worked 2.5 days per week for 2 years and coordinated a multifaceted intervention aimed at optimizing drug therapy to improve patient outcomes (blood pressure, cholesterol, diabetes, pain control, constipation, etc.) The integrated pharmacist conducted patient assessments for medication problems, optimized office system medication management (e.g. develop process for handling of medication samples), and provided education (academic detailing ) focussed on key therapeutic areas. Pharmacists were provided with ongoing support from a training and mentorship program and the services of the Ontario Pharmacists' Association Drug Information Centre.

The family physicians and other members of the practice worked closely with the pharmacist in implementing these strategic interventions. Family physicians from a range of practice models (Ontario Family Health Networks, Primary Care Networks, and other types of family physician group practices) participated in this project.

Quantitative and qualitative methods were used to evaluate the process of integration, pharmacist service uptake, drug-related patient outcomes, and the costs associated with program implementation for sustainability. The integration of the physicians and pharmacists at the practice sites were evaluated with the aim of generating a practical and transferable practice model. The main hypothesis was that pharmacist integration into family practice will optimize medication use, clinical care and clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

65 + years and any two of the following:

* Elevated blood pressure
* Elevated hemoglobin A1C
* Elevated LDL-C
* Diagnosis of hypertension and no blood pressure readings in past 12 months
* Diagnosis of diabetes and no hemoglobin A1C readings in past 12 months
* Diagnosis of hyperlipidemia and no cholesterol readings in past 12 months
* Diagnosis of osteoarthritis or rheumatoid arthritis
* Using narcotics
* Diagnosis of hypertension, diagnosis of diabetes and not using an ACE inhibitor
* Diagnosis of hypertension, elevated blood pressure and using an NSAID
* Diagnosis of hyperlipidemia, elevate dLDL-C and not using a lipid lowering agent
* Diagnosis of hypertension, high blood pressure and not using a potassium wasting diuretic

Exclusion Criteria:

* Less than one visit to family physician in past 12 months
* More than 20 visits to family physician in past 12 months
* Awaiting placement to a nursing home or long-term care facility
* Alcoholism
* Palliative care patient
* Family physician only sees patient as a home visit

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1400
Dates: Start 2004-02; Study Completion 2006-07

PRIMARY OUTCOMES:
Number and types of patients referred and assessed
Characterization and quantification of pharmacist activities
Numbers and types of drug-related problems identified and resolved
Medication changes made
Number of recommendations implemented
Process indicators (measurement of blood pressure, Cholesterol, hemoglobin A1C)
Surrogate clinical outcomes (values of blood pressure, Cholesterol, hemoglobin A1C)
Symptom improvement (constipation, pain)

SECONDARY OUTCOMES:
Health resource utilization
Satisfaction with service
Uptake of pharmacist recommendations
Extent of knowledge translation
Extent of collaboration
Satisfaction with integrated pharmacist program
Set up costs
Pharmacist and physician time costs
Travel cost
Space requirements
Medication costs
Health services utilization

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Dolovich, PharmD, MSc, Principal Investigator — McMaster University; Kevin Pottie, MD, Principal Investigator — University of Ottawa, Ottawa ON; Janusz Kaczorowski, PhD, Principal Investigator — McMaster University; Barbara Farrell, PharmD, Principal Investigator — Elisabeth Bruyere Research Institute, Ottawa, ON
Locations (3):
- Canada (3):
  - McMaster University, Hamilton, Ontario
  - University of Ottawa, Ottawa, Ontario
  - University of Toronto, Toronto, Ontario